CLINICAL TRIAL: NCT03769779
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Evaluation of the Benefits of FloraGLO™ Lutein on Skin Health
Brief Title: Evaluation of the Benefits of FloraGLO™ Lutein on Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4251KM0918
Record Dates: First submitted 2018-12-04; First posted 2018-12-10 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2018-12

CONDITIONS: Aging; Wrinkle; Skin Elasticity; Healthy; Hydration
MeSH Terms: interventions — Safflower Oil

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Envelopes that contain information regarding the coding of treatment and placebo will be provided to Sponsor, Site, and PI and kept in a secure location. Envelopes will be readily available for the investigator or site to open in the event that it becomes necessary to know which product a participant is taking for the sake of the participant health care. The sponsor must be notified of any unblinding by the site within 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Lutein (FloraGLO™) in safflower oil
  Interventions: Dietary Supplement: FloraGLO Lutein
- Placebo (Placebo Comparator): safflower oil
  Interventions: Dietary Supplement: Safflower Oil

INTERVENTIONS:
Dietary Supplement: FloraGLO Lutein — Lutein (FloraGLO™) in safflower oil
  Arms: Treatment
Dietary Supplement: Safflower Oil — Safflower Oil
  Arms: Placebo

SUMMARY:
Therefore, the present study is designed to contribute to the body of literature by investigating the effect of 12-weeks of lutein supplementation on multiple parameters of skin health and appearance in healthy women.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel twelve-week study of the performance of an oral test product to evaluate the effects of twelve weeks of lutein supplementation on skin health and appearance in healthy women. A seven-day washout period will precede the evaluation period. The subjects in each cohort will use consume one softgel of their assigned test product (treatment or placebo) daily in the morning with breakfast for 12 weeks. Changes in skin condition and appearance as well as blood chemistry will be assessed using results from expert visual grading, instrumental assessments, skin and blood assays and subjective questionnaire responses. Subjects will be recruited during the winter season to account for seasonal variations of skin parameters.

Evaluation points will occur pre-application (Baseline; Week 0) and after 42 and 84 days of use (D42, D84; Week 6, Week 12). Data will be collected on the following outcomes:

1. Skin Hydration 2. Skin texture/smoothness 2. Reduction of facial fine lines and wrinkles 3. Skin elasticity and firmness 4. Sagging skin, dry skin, skin tone, appearance from expert clinical grading and subjective questionnaire responses.

6. Skin hydration 7. Skin collagen 8. Skin lipid content. 9. Skin Carotenoids

ELIGIBILITY:
Inclusion Criteria:

1. Females in good health, and between the ages of 30 and 65 years old
2. Fitzpatrick Skin Type I-V
3. Mild to moderate loss of skin elasticity, wrinkles (global) and rough skin texture
4. Able to read, understand and sign an informed consent form
5. Willing and able to follow all study directions, attend study visits as scheduled and willing to accept the restrictions of the study
6. Willing and able to maintain regular diet, exercise, hydration, and sleep patterns throughout the study

Exclusion Criteria:

1. Participating in any other clinical study
2. Acute or chronic disease or medical condition
3. Unreliable or unlikely to be available for the duration of the study
4. Routine use of tanning bed(s)
5. History of abnormal response to sunshine
6. Current usage of medications with contraindication of enhancing sun exposure, or medications for skin conditions.
7. History of allergic reactions, skin sensitization and/or known allergies to cosmetic ingredients, toiletries, sunscreens, etc.
8. Immunocompromised subjects
9. Subject has a history of unconventional sleep patterns
10. Started Hormone Replacement Therapy within the last three months
11. Using oral contraception for less than three months
12. Known to be pregnant, lactating or planning to become pregnant within six months
13. Unable to communicate or cooperate with the Principal Investigator due to language problems, poor mental development, or impaired cerebral function

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Objective Skin Hydration | ANOVA including weeks 6 and 12
  Corneometer Value
Subjective Skin Hydration | ANOVA including weeks 6 and 12
  Subjective Questionnaire Visual Analog Scale

SECONDARY OUTCOMES:
Objective Skin Texture | ANOVA including weeks 6 and 12
  Expert clinical grading
Subjective Skin Texture | ANOVA including weeks 6 and 12
  Subjective Questionnaire Visual Analog Scale
Objective Facial Lines and Wrinkles | ANOVA including weeks 6 and 12
  Expert clinical grading
Subjective Facial Lines and Wrinkles | ANOVA including weeks 6 and 12
  Subjective Questionnaire Visual Analog Scale
Objective Sagging skin, dry skin, skin tone, and overall appearance | ANOVA including weeks 6 and 12
  Expert clinical grading
Subjective Sagging skin, dry skin, skin tone, and overall appearance | ANOVA including weeks 6 and 12
  Subjective Questionnaire Visual Analog Scale
Objective Skin elasticity | ANOVA including weeks 6 and 12
  Expert clinical grading
Subjective Skin elasticity | ANOVA including weeks 6 and 12
  Subjective Questionnaire Visual Analog Scale
Skin Collagen Ultrasound | ANOVA including weeks 6 and 12
  Ultrasound
Skin Collagen SIAsScope | ANOVA including weeks 6 and 12
  SIAsScope assessments
Skin Lipids | ANOVA including weeks 6 and 12
  HPLC of tape strips
Skin Carotenoids | ANOVA including weeks 6 and 12
  Total carotenoid concentration

CONTACTS AND LOCATIONS:
Locations (1):
- International Research Services, Inc., Port Chester, New York, United States

IPD SHARING:
Plan to Share IPD: No